CLINICAL TRIAL: NCT03530423
Title: Sensing Ventricular Arrhythmias by His Bundle Leads
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator Decision
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1804-20
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this trial is to determine if implantable cardiac device leads implanted in the His bundle are capable of detecting ventricular arrhythmias.

DETAILED DESCRIPTION:
During routine testing of implanted leads, the His bundle lead will be connected to a separate device with all therapies disabled. Testing will be done to see if the His bundle lead can detect ventricular arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing routine defibrillation threshold testing of a right ventricular implantable cardioverter defibrillator lead who also have previously placed His bundle lead or who are undergoing placement of a His bundle lead.

Exclusion Criteria:

* Individuals with contraindications to defibrillation threshold testing

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing routine defibrillation threshold testing of a right ventricular implantable cardioverter defibrillator lead who also have previously placed His bundle lead or who are undergoing placement of a His bundle lead.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Detection of ventricular arrhythmia from His bundle | 1 hour
  During defibrillation threshold testing a lead from the His bundle to an external implantable cardiac device will be used to detect an arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Deshmukh, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No